CLINICAL TRIAL: NCT04219735
Title: Effect of Minocycline on Delirium Incidence in Critically Ill Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade do Extremo Sul Catarinense - Unidade Academica de Ciecias da Saude (Other)
Responsible Party: Principal Investigator, Felipe Dal Pizzol, Head, Intensive Care Unit, São José Hospital. Head, Pathophysiology Laboratory, Universidade do Extremo Sul Catarinense, Universidade do Extremo Sul Catarinense - Unidade Academica de Ciecias da Saude
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MinoDelirium
Record Dates: First submitted 2019-10-29; First posted 2020-01-07 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Delirium; Coma
Keywords: delirium; minocycline; intensive care unit
MeSH Terms: conditions — Delirium; Coma; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Intervention Model Description: Placebo vs minocycline
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo capsules looking identical to minocycline capsules
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minocycline (Experimental): Minocycline 100 mg BID
  Interventions: Drug: Minocycline
- Placebo (Placebo Comparator): Placebo capsules identical to experimental arm
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Minocycline — Minocycline 100mg BID
  Arms: Minocycline
Drug: Placebos — Placebo
  Arms: Placebo

SUMMARY:
Delirium is a disorder of consciousness characterized by an acute onset and fluctuating course of impaired cognitive functioning. It is associated with unfavorable outcomes in hospitalized patients, including longer hospital length of stay, need for subsequent institutionalization and higher mortality rates. Patients in the intensive care unit (ICU) under mechanical ventilation and older age are at higher risk for the development of delirium. Several studies suggest that minocycline, through its anti-inflammatory effect, was able to prevent neuronal dysfunction in different models of ICU-related diseases. Thus, the present study aimed to evaluate the effect of minocycline on delirium development in critically ill patients. Patients will be randomized into one of two groups: the intervention group that will receive 100mg of minocycline 2 times a day and the placebo group. Medication or placebo will be continued for 28 days or until ICU discharge (whichever occurs first). Delirium will be diagnosed by the CAM-ICU. Coma will be defined by the Richmond Agitation-Sedation Scale (RASS) score of -4 or -5 and biomarkers will be used as alternative outcomes related to the pathophysiology of the disease (IL-1, IL-6, IL-10, and BDNF).

ELIGIBILITY:
Inclusion Criteria:

* Clinical or surgical patients,
* Over 18 years,
* Expected ICU stay of at least 2 days estimated by the attending intensivist,
* Agree to participate in the study

Exclusion Criteria:

* Delirium prior to inclusion,
* Diagnosis of Parkinson's disease
* Diagnosis of dementia,
* Alcohol abuse history,
* Acute neurological condition at admission
* History of psychiatric disease
* Use of antipsychotics
* Pregnant or breastfeeding women,
* Expectation of death within 2 days
* Hospitalized for exclusive palliative care
* Known allergy to minocycline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Delirium and subsyndromal delirium incidence during ICU stay | up to 28 days
  Number of patients with delirium

SECONDARY OUTCOMES:
Days in delirium during ICU stay | up to 28 days
  Number of days being in delirium
Coma-delirium free days during ICU stay | up to 28 days
  Number of days free of coma or delirium
Length of mechanical ventilation during ICU stay | up to 28 days
  Number of days in mechanical ventilation
Length of ICU stay | up to 28 days
  Number of days in the ICU
ICU mortality | up to 28 days
  Number of dead during ICU stay
Hospital mortality | up to 90 days
  Number of dead during hospital stay
Long-term quality of life measured by the 12-Item Short-Form Health Survey V2 | until 12 months after hospital discharge
  Quality of life measured after hospital discharge
Long-term cognitive dysfunction measured by Montreal Cognitive Assessment score | until 12 months after hospital discharge
  Cognitive function after hospital discharge
Plasma levels of interleukin-6, interleukin-10, brain derived neural factor and S100-B | At Day 1 and 3 of ICU stay, and hospital discharge
  Inflammatory and brain derived plasma biomarker levels
Long-term Post-Traumatic Stress Disorder measured by Impact of Event Scale-Revised | until 12 months after hospital discharge
  Post-Traumatic Stress Disorder symptoms after hospital discharge measured by the Impact of Event Scale-Revised ranging from 0 to 88, higher values indicate more severe symptoms
Long-term depression and anxiety symptoms measured by Hospital Anxiety and Depression Scale | until 12 months after hospital discharge
  Depression and anxiety symptoms after hospital discharge measured by Hospital Anxiety and Depression Scale, ranging from 0 to 21, higher values indicate more severe symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- São José Hospital, Criciúma, Santa Catarina, Brazil

REFERENCES:
- [Derived] Dal-Pizzol F, Coelho A, Simon CS, Michels M, Corneo E, Jeremias A, Damasio D, Ritter C. Prophylactic Minocycline for Delirium in Critically Ill Patients: A Randomized Controlled Trial. Chest. 2024 May;165(5):1129-1138. doi: 10.1016/j.chest.2023.11.041. Epub 2023 Dec 1. PMID 38043911